CLINICAL TRIAL: NCT04954963
Title: Objective to Explore the Clinical Application Value of Spectral CT Mar Technology and Magnetic Resonance Mavric, Semac Sequence in Removing Artifacts of Orthopedic Metal Internal Fixation
Brief Title: CT Mar Technology and MR Mavric, Semac Sequence in Removing Artifacts of Orthopedic Metal Internal Fixation
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019317
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2019-12

CONDITIONS: Spinal Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conventional examination: patients undergo conventional examination
- Reduce metal artifacts examination: patients undergo reduce metal artifacts examination
  Interventions: Diagnostic Test: Reduce metal artifacts examination

INTERVENTIONS:
Diagnostic Test: Reduce metal artifacts examination — patients undergo reduce metal artifacts examination
  Groups: Reduce metal artifacts examination

SUMMARY:
1. Objective to compare the effect of single energy imaging and mar technology in reducing artifacts of knee and hip replacement, and to explore the appropriate keV range of Mar technology in removing metal artifacts.,2. Objective to compare the effects of different MRI sequences (mavric / semac, stir, ideal, FSE) in removing artifacts of spinal internal fixation, knee and hip replacement.

DETAILED DESCRIPTION:
Conventional spiral CT [4] examination will form black-and-white stripe artifacts around the metal implant, making the display of adjacent important structures unclear. In routine MRI examination [5], metal will interfere with the uniformity of local magnetic field, resulting in signal loss, and the artifacts will seriously affect the observation of bone and its surrounding structures.

The purpose of this study was to comprehensively evaluate the effect of Mar technology on reducing metal artifacts after internal fixation and joint replacement, and then to explore the appropriate keV range of Mar technology to reduce metal artifacts. We also aim to compare the reduction effect of different sequences of MRI on internal fixation artifacts after internal fixation and joint replacement, and to explore the sequence suitable for clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients after spinal internal fixation or knee or hip replacement

Exclusion Criteria:

* Patients with poor image quality caused by their own factors such as patients' movement can not meet the diagnostic requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From December 2019 to October 2020, patients who were reexamined after spinal internal fixation or knee and hip replacement in Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Artifact index | 2020.10.15-2020.10.30
  AI in region of interest

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Yuan, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China